CLINICAL TRIAL: NCT05925452
Title: A Multicenter, Randomized Phase II/III Clinical Study to Evaluate the Efficacy and Safety of GenaKumab in the Treatment of Active Systemic Juvenile Idiopathic Arthritis.
Brief Title: To Evaluate the Efficacy and Safety of Genalumab for Injection in the Treatment of Active Systemic Juvenile Idiopathic Arthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci048-201
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Active Systemic Juvenile Idiopathic Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GenaKumab (Experimental): 15 subjects: GenaKumab 3.0mg/kg dose group and 4.0 mg/kg dose group, Subcutaneous injection, Q4w
  Interventions: Drug: GenaKumab

INTERVENTIONS:
Drug: GenaKumab — GenaKumab 3.0mg/kg dose group : GenaKumab 3.0 mg/kg, Subcutaneous injection, Q4w； GenaKumab 4.0 mg/kg dose group : GenaKumab 4.0 mg/kg, Subcutaneous injection, Q4w

SUMMARY:
A multicenter, randomized Phase II/III clinical study to evaluate the efficacy and safety of GenaKumab in the treatment of active systemic juvenile idiopathic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, with the remaining before age 2 years old or more and & lt; 18 years old;
* 2001 ILAR classification criteria for the diagnosis of confirmed sJIA 2 or more months: onset age must & lt; At 16 years of age, symptoms included: ≥1 case of arthritis, accompanied by or prior to ≥2 weeks of recurrent fever, including remittenor fever for ≥3 consecutive days (maximum daily body temperature ≥39 ° C, body temperature falling below 37 ° C between 2 heat peaks), accompanied by at least one of the following symptoms: ① a transient, non-fixed erythematous rash; ② systemic lymph node enlargement; Swelling of the liver and/or spleen; ④ Serositis.
* Agree to use effective means of contraception throughout the study period and for 6 months after the end of treatment.

Exclusion Criteria:

* Pregnant or lactating female subjects
* A history of allergic reactions to investigational drugs or to molecules with similar structures; Those who cannot be given intramuscular injections；
* History of pericarditis, myocarditis, serositis, bacterial heart valve or endocarditis within 6 months before screening; Patients who had been diagnosed with MAS within 6 months prior to screening, or had relevant symptoms and signs at screening, and were suspected of having MAS as assessed by the investigators；
* There are other rheumatic diseases such as Kawasaki disease, polyarteritis nodosa and so on. History of autoinflammatory diseases such as familial Mediterranean fever, high IgD syndrome, NLRP3-related autoinflammatory diseases；
* Patients with a history of interstitial lung disease, pulmonary fibrosis, alveolar proteinosis, or pulmonary hypertension; Patients with a history of repeated invasive fungal infection; In the 7 days prior to randomization, there were infections that required control with systemic antigenic microbiotics (including antibacterial, antiviral, antifungal, etc.)；
* Subjects with a history of TB exposure or suspected TB symptoms.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 221 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-03-24 (Estimated); Study Completion 2028-06-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with successful glucocorticoid reduction by the end of the treatment period | 24 Week

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Children's Hospital Affiliated to Capital Medical University, Beijing, Benjing
  - Children's Hospital Affiliated to Chongqing Medical University, Chongqing, Chongqing Municipality
  - Hunan Children's Hospital, Changsha, Hunan
  - Children's Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Pediatric Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Xi'an Children's Hospital, Xi’an, Shanxi
  - Chengdu Women and Children's Central Hospital, Chengdu, Sichuan
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang